CLINICAL TRIAL: NCT03127761
Title: Assessment of Allogeneic Hematopoietic Cell Transplantation in Medicare Beneficiaries With Multiple Myeloma: A Study to Develop Evidence of Effectiveness for the Centers for Medicare and Medicaid Services (CMS)
Brief Title: Assessment of Allogeneic Hematopoietic Cell Transplantation in Medicare Beneficiaries With Multiple Myeloma
Status: Recruiting | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Other Study IDs: 17-CMS-MM
Record Dates: First submitted 2017-04-18; First posted 2017-04-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allogeneic HCT: Prospectively enrolled cohort of patients receiving allogeneic hematopoietic cell transplantation for multiple myeloma
  Interventions: Other: Allogeneic Hematopoietic Stem Cell Transplant
- Historical autoHCT: Historical cohort of patients with autologous hematopoietic cell transplantation between 2010 and 2016

INTERVENTIONS:
Other: Allogeneic Hematopoietic Stem Cell Transplant — This observational study will compare outcomes of prospectively enrolled HCT recipients with outcomes of a cohort of matched autoHCT controls.
  Groups: Allogeneic HCT

SUMMARY:
Multiple myeloma (MM) is the second most common hematologic malignancy in adults. The current standard of care for MM patients fit to undergo high dose conditioning chemotherapy is an autologous HCT (autoHCT). Allogeneic HCT (alloHCT) is the only potentially curative therapy available to patients with MM. However, the significant morbidity and mortality of this procedure historically limited its application in older patients.

Thus, although potentially curative, standard risk MM patients have excellent prognoses in the era of novel therapies which reduces the overall benefit of alloHCT. However, because the outcomes for high-risk MM remain poor despite the best available standard therapies (overall survival of 24-36 months), initial data suggest that alloHCT should be explored in this subset.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is the second most common hematologic malignancy in adults. Overall survival (OS) in MM has improved significantly in the last 15 years with the emergence of novel therapies such as thalidomide, bortezomib and lenalidomide. The median life expectancy of patients with MM treated in the current era is more than 6 years, while SEER data from a slightly earlier time period (2008-12) estimated the 5 year survival at 48.5%. However, prognosis is not uniform and varies considerably based on a presenting features and response to therapy.

The current standard of care for MM patients fit to undergo high dose conditioning chemotherapy is an autologous HCT (autoHCT). There is controversy regarding the timing of autoHCT after initial novel therapy induction with randomized trials showing similar OS whether done early or delayed to time of relapse as salvage therapy. However, more recent trials comparing early versus delayed transplant support the benefit of early upfront autoHCT.

Allogeneic HCT (alloHCT) is the only potentially curative therapy available to patients with MM. However, the significant morbidity and mortality of this procedure historically limited its application in older patients. Current data from the Center for International Blood and Marrow Research (CIBMTR) show transplant-related mortality rates of 23 (20-26)% at 5 years with myeloablative conditioning.

Thus, although potentially curative, standard risk MM patients have excellent prognoses in the era of novel therapies which reduces the overall benefit of alloHCT. However, because the outcomes for high-risk MM remain poor despite the best available standard therapies (overall survival of 24-36 months), initial data suggest that alloHCT should be explored in this subset.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiary
* Stage II or III multiple myeloma and/or primary plasma cell leukemia
* Eligible to receive an allogeneic HCT from any suitable allogeneic donor (as determined by the transplant center) including umbilical cord blood
* Will receive allogeneic HCT at a US transplant center
* Agree to submit comprehensive clinical data on their pre- and post-transplant clinical status and outcomes to the CIBMTR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A prospective cohort study of approximately 544 patients receiving allogeneic HCT for multiple myeloma in CIBMTR centers in the US matched to a historical control patients treated with autoHCT between 2010 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 544 (Estimated)
Dates: Start 2017-07-25 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Compare five-year survival | 5 years post transplant
  Compare five-year overall survival between the alloHCT cohort and an age and disease risk matched cohort of autoHCT patients

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 years post transplant
  five-year PFS probabilities between the AlloHCT cohort and an age and disease risk matched cohort of autoHCT patients
Relapse or progression | 5 years post transplant
  Myeloma recurrence or progression will be defined per International Myeloma Working Group (IMWG) guidelines
Transplant related mortality | 5 years post transplant
  Death from any cause within 28 days after alloHCT or death in the absence of progression/relapse of MM after day 28 post transplant
Incidence of acute GVHD | 5 years post transplant
  Occurrence of Grade I, II and III/IV skin, gastrointestinal, or liver abnormalities fulfilling the Consensus criteria of Grades II-IV acute GVHD
Incidence of chronic GVHD | 5 years post transplant
  Occurrence of symptoms in any organ system fulfilling the criteria of chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Anita D'Souza, MD, MS, Study Chair — CIBMTR, Medical College of Wisconsin; Parameswaran Hari, MD, MS, Study Chair — CIBMTR, Medical College of Wisconsin
Locations (1):
- Center for International Blood and Marrow Transplant Research, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided